CLINICAL TRIAL: NCT04622657
Title: Validity Reliability of The Dubousset Functional Test in Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Ayşe Abit Kocaman, Principal Investigator, Kırıkkale University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Parkinson Disease Assesment
Record Dates: First submitted 2020-10-29; First posted 2020-11-10 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Parkinson Disease; Balance; Distorted; Fall; Gait Disorders, Neurologic
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- parkinson disease (Experimental): Assessment
  Interventions: Other: dubousset functional test

INTERVENTIONS:
Other: dubousset functional test — Dubousset Function Test, 3-m backwards walk test, timed up and go test,Tinnetti Balance and Gait Test, Berg BalanceTest, Functional Reach Test

SUMMARY:
In order to achieve collaborative patient-centered rehabilitation in Parkinson's disease, detailed evaluation of walking and balance in evaluating the perceived difficulty in daily life is important to evaluate the progression of the disease and its response to treatments.

In the literature, there are many scales that evaluate balance and functional performance in Parkinson Disease. However there is no validity and reliability study of Dubousset Function Test developed to evaluate balance and functional performance of Parkinson Disease. For this reason, the aim of study is to examine the validity and reliability of Dubousset Function Test in Parkinson Disease.

DETAILED DESCRIPTION:
Balance disorders are very common in patients with Parkinson's, and these disorders significantly affect the patient's body alignment and participation. Especially during walking, balance disorders occur, resulting in falls, disability and injury in the advanced stage of the disease. As a result of these losses in patients, falls can be seen, and the severity of disability that increases with age affects the quality of life of individuals by affecting their living in their own homes.

Dubousset Functional Test (DFT); A conceptually practical four-component assessment test has been proposed by Dr. Jean Dubousset to assess the functional capacity of adult individuals. The validity of the test was made in individuals with spinal deformity. DFT; It consists of four components: getting up from a chair without arms and walking 5 meters forward and backward, descending and climbing steps, transition from standing to sitting on the ground, and the dual task test in which the individual walks while counting down from 50 at the same time

In the literature, there are many scales that evaluate balance and functional performance in Parkinson Disease. However there is no validity and reliability study of Dubousset Function Test developed to evaluate balance and functional performance of Parkinson Disease. For this reason, the aim of study is to examine the validity and reliability of Dubousset Function Test in Parkinson Disease.

ELIGIBILITY:
Inclusion Criteria:

Being diagnosed with Parkinson's Disease (Hoehn Yahr level (1-3)

* Volunteering to participate in research and approving the informed consent form Being over the age of 40
* Using stable Parkinson's Disease medication for at least 4 weeks
* No cooperation and communication problems

Exclusion Criteria:

* • Individuals with any other neurological and orthopedic problems Uncontrollable hypertension To your serious disk Significant comorbidity affecting balance and gait

  * Those with cooperation and communication problems

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-25 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Dubousset Function Test | through study completion, an average of 1 year
  The four components of the DFT included (1) the Up Walking Test: participants rose without assistance from a and seated position in a chair that did not have arms, walked 5 meters (500 cm) forward before stopping, walked backwards 5 meters, and sat again without assistance; (2) the Steps Test: from a starting position 50 cm away, volunteers climbed three stairs, turned around on the third step (top), and walked down the three steps; (3) Down and Sitting Test: from a standing position, participants sat on the ground and stood up again, using assistance as needed; (4) Dual-Tasking Test: participants walked 5 meters forward, turned around, and walked 5 meters back to the starting position while performing a working memory test (counting down from 50 by intervals of 2).
timed up and go test | through study completion, an average of 1 year
  A standard chair is used for testing. First, the patient is asked to sit on the chair. The patient is then asked to stand up and walk regularly at a distance of 3 meters with a predetermined length, then return to the chair after 3 meters.
3-m backwards walk test | through study completion, an average of 1 year
  A distance of 3 m is measured and marked with black tape. Individuals are asked to follow the heel and black band.
  With the 'start' command they are asked to walk backwards quickly. When the distance of 3 m is completed, a stop is instructed. Individuals are not allowed to run during the test. They are allowed to look back if they wish. The assessor walks behind individuals throughout the test. The test is repeated 3 times, the averages are recorded
Tinetti Balance and Gait Test | through study completion, an average of 1 year
  In the test used to evaluate balance, walking score is maximum 12 points, balance score is maximum 16 points and a total of 28 points.
Funtional Reach Test | through study completion, an average of 1 year
  It is used to measure both the balance of the individual functionally and the amount of dynamic reach It is used to measure both the balance of the individual functionally and the amount of dynamic reach
Berg Balance Test | through study completion, an average of 1 year
  The BBS consists of 14 items to directly monitor the maintenance of body balance during performance

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Abit Kocaman, PhD, Principal Investigator — Kırıkkale University
Locations (1):
- Ayşe Abit Kocaman, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diebo BG, Challier V, Shah NV, Kim D, Murray DP, Kelly JJ, Lafage R, Paulino CB, Passias PG, Schwab FJ, Lafage V. The Dubousset Functional Test is a Novel Assessment of Physical Function and Balance. Clin Orthop Relat Res. 2019 Oct;477(10):2307-2315. doi: 10.1097/CORR.0000000000000820. PMID 31135543